CLINICAL TRIAL: NCT01325974
Title: Time to Become Negative of Three Rapid Diagnostic Tests for Malaria in Children Under 5 Years of Age. Evaluation in Two Different Malaria Epidemiological Settings in Greater Mbarara District, South Western Uganda
Brief Title: Time to Become Negative of Three Rapid Diagnostic Tests for Malaria
Status: Completed | Type: Observational
Sponsor: Epicentre (Other)
Collaborators: Medecins Sans Frontieres, Netherlands (Other)
Responsible Party: Sponsor
Other Study IDs: Epicentre/Mba/2011/TTBN-RDTmal
Record Dates: First submitted 2011-03-29; First posted 2011-03-30 (Estimated); Last update posted 2015-11-30 (Estimated); Status verified 2015-11

CONDITIONS: Malaria, Falciparum
Keywords: Malaria; Plasmodium falciparum; Diagnosis; Rapid diagnostic test; malaria transmission
MeSH Terms: conditions — Malaria, Falciparum; Malaria; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood smears for microcopy
Oversight: Data Monitoring Committee: No

SUMMARY:
Background: Antigen-detecting rapid diagnostic tests (RDTs) for malaria provide the possibility of a parasite-based diagnosis in areas where good quality microscopy can not be achieved.

P. falciparum tests targeting the histidine-rich protein (HRP2) antigen are generally more sensitive than tests targeting the Plasmodium lactate dehydrogenase (pLDH) antigen. However, as the HRP2 antigen is eliminated from the bloodstream more slowly than the pLDH antigen, HRP2-based tests can give a positive result two weeks or more after the patient has taken an effective treatment, while pLDH tests generally turn negative a few days after. The use of an RDT positive result in a routine patient care is therefore challenged by the interpretation of whether the result is due to a lasting effect of the already treated infection or to a new infection. The interpretation might also be affected by the level of malaria transmission in the area.

Objective: The objective of this study is to estimate the proportion of positive tests in patients successfully treated for malaria (smear negative) at different time points in time after treatment, for three rapid diagnostic tests: SD Bioline Malaria Antigen P.f. (catalogue number: 05FK50-02-4), CareStart Malaria HRP2 (Pf) (catalogue number: G0141) and CareStart Malaria pLDH (PAN) (catalogue number: G0111). The study will be carried out in two settings with known low and high malaria transmission levels in order to provide guidance of interpretation of a RDT positive result depending on the intensity of malaria transmission.

Secondary objectives will be to measure the sensitivity and specificity of the malaria rapid tests compared to smear microscopy, to estimate the median time to become negative for each of the tests and to estimate the proportion of positive tests and the median time to become negative according to the initial parasitaemia and the presence of gametocytes.

DETAILED DESCRIPTION:
The study population will be patients under 5 years of age who attend the consultation service of one health centre of Mbarara municipality (low transmission setting) and one health centre in Kazo sub-county (high transmission setting) and for whom the clinical diagnosis of malaria is confirmed by smear microscopy and with at least one positive RDT. Patients with general signs of danger of severe malaria or who took a full course of antimalarial treatment in the previous 2 weeks will be excluded. Written consent will be sought from all participants.

A total of 212 patients will be included in each setting. The sample size was based of a minimum accuracy of 8% around a proportion of 50% positive RDTs to which a 15% was added for patients who will not be positive for all RDTs or will be secondarily excluded from the analysis.

A three-day artemether-lumefantrine will be given to enrolled cases and treatment intake will be supervised. RDTs and a blood smear microscopy will be repeated at day 2, 3, 5, 7, 14, 21, 28, 35 and 42 after inclusion until all RDTs become negative. Follow-up will not last longer than 42 days.

The proportion and 95% confidence intervals of positive tests among patients with a negative thick smear will be calculated for each day of follow-up. Moreover the investigators will identify for each test a regression model to estimate the number of days required to obtain a 50, 25, 10 and 5% probability of having a false positive RDT result.

Sensitivity, specificity, positive and negative predictive values will be estimated for each RDT independently using the result of microscopy as a reference. The analysis will be performed using the day 0 results for all patients enrolled in the study.

ELIGIBILITY:
Inclusion Criteria (sensitivity/specificity analysis):

* Age under 5 years
* Clinical malaria defined as fever (axillary temperature ≥ 37.5°C) or history of fever in the previous 48 hours
* Weight ≥ 5 kg
* Informed consent given by the parent or a tutor

Additional inclusion criteria (time to become negative analysis):

* Positive blood smear with a Plasmodium falciparum monoinfection at the day of inclusion
* At least one RDT positive at the day of inclusion
* High probability of coming to all follow-up visits

Exclusion Criteria (time to become negative analysis):

* General signs of danger or of severe malaria according to the WHO criteria
* Treatment course of antimalarials in the previous 2 weeks

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population will be patients under 5 years of age who attend the consultation service of one health centre of Mbarara municipality (low transmission setting) and one health centre in Kazo sub-county (high transmission setting).
Sampling Method: Non-Probability Sample
Enrollment: 424 (Actual)
Dates: Start 2011-09; Primary Completion 2013-02 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
To estimate the proportion of positive tests in patients successfully treated for malaria (smear negative) at different time points after treatment, for three rapid diagnostic tests: two HRP2 test and one pLDH test. | day 2, 3, 5, 7, 14, 21, 28, 35 and 42 after the start of antimalarial treatment intake

SECONDARY OUTCOMES:
To measure the sensitivity and specificity of the malaria rapid tests compared to smear microscopy. | The day of patient's enrollment only (day 0)
To estimate the median time to become negative for each of the rapid diagnostic test. | day 2, 3, 5, 7, 14, 21, 28, 35 and 42 after the start of antimalarial treatment intake
To estimate the proportion of positive tests among smear negative results and the median time to become negative according to the initial parasitaemia and the presence of gametocytes. | day 2, 3, 5, 7, 14, 21, 28, 35 and 42 after the start of antimalarial treatment intake

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Grandesso, MSc, Principal Investigator — Epicentre; Carolyn Nabasumba, MD, Study Chair — Epicentre; Yap Boom, MSc, PhD, Study Chair — Epicentre; Anne-Laure Page, PhD, Study Chair — Epicentre; Mathieu Bastard, MSc, Study Chair — Epicentre; Jean-François Etard, MD, PhD, Study Director — Epicentre
Locations (2):
- Uganda (2):
  - Kazo level 4 health centre, Kazo, Greater Mbarara District
  - Mbarara Municipality level 2 health centre, Mbarara, Greater Mbarara District

REFERENCES:
- [Derived] Grandesso F, Nabasumba C, Nyehangane D, Page AL, Bastard M, De Smet M, Boum Y, Etard JF. Performance and time to become negative after treatment of three malaria rapid diagnostic tests in low and high malaria transmission settings. Malar J. 2016 Oct 4;15(1):496. doi: 10.1186/s12936-016-1529-6. PMID 27716244